CLINICAL TRIAL: NCT05626647
Title: Etiology of Anemia Among Preschool Children and Its Public Health Implication in Selected Regions of Ethiopia: A Community-Based Longitudinal Study
Brief Title: Etiology of Anemia Among Preschool Children in Ethiopia
Status: Completed | Type: Observational
Sponsor: Oklahoma State University (Other)
Collaborators: Ethiopian Public Health Institute (Other Government); Addis Ababa University (Other)
Responsible Party: Principal Investigator, Solomon Hailu, Principal Investigator, Oklahoma State University
Other Study IDs: IRB-21-505
Record Dates: First submitted 2022-11-15; First posted 2022-11-25 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Anemia
Keywords: Etiology; Anemia; Preschool
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Biospecimen Retention: Samples With DNA — The hemoglobinopathies test will be performed to assess the genetic alteration of the individual hemoglobin synthesis status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to determine the etiology of anemia among preschool children in selected regions of Ethiopia. The study is a longitudinal observational study to assess the determinant factors of anemia in two different seasons.

The main questions it aims to answer are:

1. What is the prevalence and etiology of anemia in the two different (Post and Pre-harvest) seasons?
2. What is the strength of the interaction between anemia and each of the determinant factors being considered?

The participant's dietary intake and anthropometric measurement have been assessed, and biological samples (Blood and Stool) were collected to determine the prevalence of anemia and the factors contributing to it.

DETAILED DESCRIPTION:
Background: Although the country made a significant change in the burden of malnutrition in all its forms in the past two decades, the issue remains unacceptably high across all regions of Ethiopia. The national prevalence of anemia among children 6-59 months was very high 57% and one of the public health concerns in 2016. Although the country is known as a data-rich country, in some specific indicators, there is a lack of data and evidence to alleviate the nutritional gaps through an informed decision-making process. In this particular case, there is a lack of evidence relating to child anemia in Ethiopia, especially since there is no comprehensive information about the determinant factors of anemia.

Objective: The objective of the current survey is to determine the etiology of anemia and its public health implications among under-five children in selected ecological zones of Ethiopia at different seasons.

Method: This survey will be a community-based, longitudinal panel study and will be conducted in two different (post-harvest and pre-harvest) seasons in the 2014 Ethiopian calendar year. A nationally representative sample was calculated and allocated to three purposely selected regions (Amhara, Southern Nation, Nationalities, and Peoples' Region (SNNPR), and Somali) in consideration of three different ecological zones (lowlands, midlands, and highlands). The study population will be children aged 6 - 59 months with caregivers/mothers with a sample size of 1212 under-five children from 1212 households. The indicators collected for the survey are dietary intake, anthropometric measurement, and biological samples (Blood and Stool).

Expected benefit: The findings of this survey will provide information on the etiology of anemia that will inform short-term policy decisions, especially for case-specific nutrition-sensitive interventions, and that will contribute to long-term policy decisions for comprehensive nutrition intervention programs.

ELIGIBILITY:
Inclusion Criteria:

* Children 6-53 months during the baseline survey and who have stayed more than 6 months in the selected household of the Amhara or SNNPR or Somali regions of Ethiopia and have no plan to move from the study area during the study period

Exclusion Criteria:

* Children older than the youngest child between 6-53 months of age (If more than one eligible child is in the Household) during the baseline survey.
* Children with severe illness
* Guests
* If participants lose their willingness to participate in this study

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children at the age of 6 to 59 months in each randomly selected eligible household of the Amhara or SNNPR or Somali regions of Ethiopia were the study population for this study but, during the baseline survey, we found children 6 to 53 months to retain the same child at the endline survey below five years old.
Sampling Method: Probability Sample
Enrollment: 590 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-09-04 (Actual)

PRIMARY OUTCOMES:
Prevalence of anemia among preschool children in selected regions of Ethiopia in the two different (Post and Pre harvest) seasons? | From November 2021 to September 2022
  Blood hemoglobin level below 11mg/dL

SECONDARY OUTCOMES:
Factors contributing to anemia anemia among preschool children in selected regions of Ethiopia in the two different (Post and Pre harvest) seasons? | From November 2021 to September 2022
  Micronutrient deficiency, presence of infectious disease, and genetic problems contributing to low hemoglobin concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Stocker, Prof, Study Chair — Oklahoma State University
Locations (1):
- Ethiopian Public Health Institute, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data (IPD) can be shared upon request and signing of an agreement between the Ethiopian Public Health Institute and the interested party.

REFERENCES:
- [Result] Anemia prevalence among preschool children in 2016 is 57%. EDHS, "Ethiopian Demography and Health Survey 2016, Central Statistical Agency (CSA).," Addis Ababa, Ethiopia, 2016.